CLINICAL TRIAL: NCT03334812
Title: A Randomized, Placebo-controlled, Patient and Investigator Blinded, Single Dose, Proof of Concept Study Investigating the Safety, Tolerability and Preliminary Efficacy of Intra-articular LNA043 in Regenerating the Articular Cartilage of the Knee at Donor Sites in Patients Undergoing Autologous Chondrocyte Implantation
Brief Title: Study on Safety, Tolerability and Prelimenary Efficacy of LNA043 in Patients Undergoing Autologous Chondrocyte Implantation
Acronym: ACI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early based on an interim analysis of 14 subjects, which demonstrated a favorable safety and tolerability profile.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNA043X2201
Record Dates: First submitted 2017-10-16; First posted 2017-11-07 (Actual); Results first posted 2020-04-17 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Knee Cartilage Lesion
Keywords: cartilage lesion, ACI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LNA043 20mg/ml (Experimental): LNA043 20mg/ml single dose
  Interventions: Biological: LNA043
- Matching placebo to 20mg (Placebo Comparator): Matching placebo to 20mg/3ml, single dose
  Interventions: Biological: placebo to LNA043
- LNA043 40mg/ml (Experimental): LNA043 40mg/ml single dose
  Interventions: Biological: LNA043
- Matching placebo to 40mg (Placebo Comparator): Matching placebo to 40mg/4ml, single dose
  Interventions: Biological: placebo to LNA043

INTERVENTIONS:
Biological: LNA043 — LNA043 Single dose
  Arms: LNA043 20mg/ml; LNA043 40mg/ml
Biological: placebo to LNA043 — placebo to LNA043 single dose
  Arms: Matching placebo to 20mg; Matching placebo to 40mg

SUMMARY:
The purpose of this study was to assess safety, tolerability, pharmacokinetics and preliminary efficacy of a single intra-articular (i.a.) administration of LNA043 in regenerating the articular cartilage of the knee, in a standardized clinical scenario of acute cartilage defect. The study aimed at characterizing the mechanism of action of LNA043

DETAILED DESCRIPTION:
This was a non-confirmatory, patient and investigator blinded, randomized, placebo-controlled, parallel group, single dose study in patients with cartilage lesions undergoing autologous cartilage implantation (ACI). Participants were treated only on one occasion (Day 1) with a single i.a. injection that was performed under arthroscopic visualization and followed up for 28 weeks.

Originally approximately 22 patients were planned to be enrolled in two cohorts (LNA043 20 mg and LNA043 40 mg). The study was terminated before any patient was randomized into the LNA043 40 mg cohort

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Patient is ≥18 and≤ 50 years old at time of screening
* Patient has a body mass index (BMI) <30 kg/m2 at screening
* Patient has a localized articular cartilage defect of the knee and is scheduled for an ACI procedure
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* Patient has radiologically apparent degenerative joint disease in the target knee as determined by Kellgren and Lawrence grade ≥2 based on X-ray evaluation performed within 6 months from screening
* Patient has unstable knee joint or insufficiently reconstructed ligaments, based on medical history and physical examination by the investigator.
* Patient scheduled for a concomitant articular surgical procedure (e.g., anterior cruciate ligament reconstruction) other than debridement or partial meniscectomy
* Patient has malalignment (valgus- or varus-deformity) in the target knee ≥ 5° based on based on X-ray evaluation performed within 6 months from screening.at screeningmedical history. In suspected cases, the mechanical axis must be established radiographically through complete leg imaging during standing and in postero-anterior projection.
* Patient has a known autoimmune disease, inflammatory arthropathy (including but not limited to rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, CPPD, gout), active acute or chronic infection of the joint, recent Lyme disease to the knee, systemic cartilage disorder, or a known systemic connective tissue disease.
* Patient has had surgical treatment of the target knee using autologous osteochondral transplantation/mosaicplasty within 12 months prior to screening (Note: prior diagnostic arthroscopy with debridement and lavage, meniscal surgery, microfracture, anterior cruciate ligament reconstruction, and extra-articular surgery e.g., high-tibial osteotomy are acceptable).
* Patient is unable to undergo magnetic resonance imaging (MRI) or presents absolute contraindications to MRI (e.g., metallic implants, metallic foreign bodies, pacemaker, defibrillator).
* Patient taking medications prohibited by the protocol: corticosteroids by any route (except topical) from 4 weeks prior to screening; nonsteroidal anti-inflammatories or aspirin (greater than 100 mg per day) within 2 weeks prior to screening; paracetamol greater than 3000 mg per day within 2 weeks prior to screening; glucosamine or chondroitin sulfate within 2 weeks prior to screening; any local treatment i.a. into the knee within 3 months from screening.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 15 days after stopping of investigational drug.
* Regular smokers (use of tobacco/nicotine products in the previous 3 months > 5 cigarettes/day). Urine cotinine levels will be measured during screening for all subjects. Regular smokers will be defined as any subject who reports tobacco use of > 5 cigarettes/day and/or who has a urine cotinine ≥ 500 ng/mL.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from 3 clinical sites in Austria.
Pre-assignment Details: The original set up of this trial was for 2 cohorts of LNA043 (20 mg and 40 mg). The trial was terminated before any patient in the LNA043 40 mg cohort was randomized
Groups:
- LNA043 20mg: LNA043 20mg/3ml single dose
- LNA043 40mg: LNA043 40mg/4ml single dose
Period: Overall Study
Arm/Group | LNA043 20mg | Matching Placebo to 20mg | LNA043 40mg | Matching Placebo to 40mg
Started | 9 | 5 | 0 | 0
Completed | 9 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNA043 20mg | Matching Placebo to 20mg | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (6.16) | 39.4 (7.40) | 34.0 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 6 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in GAG Content
Description: Sodium MRI-based measurements of change from baseline in glycosaminoglycan (GAG) content were assessed from both defective sites and a nearby healthy cartilage region (as a reference tissue). Specifically, the ratio of normalized sodium signal in the surgically created defect (SCD or donor site) to healthy non-weight bearing region (HNWB), i.e. SCD/HNWB and the defect to be treated (DTBT or main lesion) to healthy weight bearing region (HWB), i.e. DTBT/HWB was of major interest
Time Frame: Baseline, Week 4
Population: Pharmacodynamic analysis set. Subjects with any available PD data, who received any study drug and experienced no protocol deviations with relevant impact on PD data.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 7 | 2
Ratio
  SCD/HNWB | 0.24 (0.06) | 0.06 (0.12)
  DTBT/HWB | 0.08 (0.04) | 0.09 (0.09)
Statistical Analysis 1: Comparison: LNA043 20mg vs Matching Placebo to 20mg; SCD/HNWB; Test type: Superiority; p = 0.1219, Mixed Effect Model Repeat Measurement; Mean Difference (Net) = 0.18, 95% CI 2-sided [-0.15 to 0.51]
Statistical Analysis 2: Comparison: LNA043 20mg vs Matching Placebo to 20mg; DTBT/HWB; Test type: Superiority; p = 0.5438, Mixed Effect Model Repeat Measurement; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.28 to 0.25]

2. Primary Outcome: Bi-layer Collagen Organization Based on MRI Measurements
Description: MRI T2 maps were generated and zonal T2 ratios (superficial layer T2 / deep layer T2) were calculated to assess the collagen fiber organization in the surgically created defect (SCD) and defect to be treated (DTBT) cartilage regions.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 7 | 4
Ratio | 1.01 (0.07) | 0.95 (0.09)
Statistical Analysis 1: Comparison: LNA043 20mg vs Matching Placebo to 20mg; Test type: Superiority; p = 0.3067, Mixed Effect Model Repeat Measurement; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.19 to 0.31]

3. Secondary Outcome: Change From Baseline in International Cartilage Repair Society (ICRS) Scoring
Description: Extent of the repair tissue at the donor site before surgery. Each criterion was evaluated based on the visual analog scale and graded from 0 (best) to 100 (worst).
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 8 | 4
Unit on a scale
  Abnormal Calcification/Ossification | 98.75 (1.05) | 100.00 (1.48)
  Cell Morphology: number analyzed (Participants) | 7 | 3
  Cell Morphology | 61.43 (14.14) | 56.67 (21.60)
  Chondrocyte clustering: number analyzed (Participants) | 7 | 3
  Chondrocyte clustering | 85.71 (8.37) | 85.00 (12.78)
  Inflammation | 92.50 (2.15) | 98.75 (3.04)
  Matrix Staining: number analyzed (Participants) | 7 | 3
  Matrix Staining | 57.14 (12.17) | 25.00 (18.59)
  Overall assessment: number analyzed (Participants) | 7 | 3
  Overall assessment | 49.29 (12.23) | 55.00 (18.68)
  Tissue Morphology: number analyzed (Participants) | 7 | 3
  Tissue Morphology | 71.43 (7.78) | 65.00 (11.88)
  Vascularisation in repaired tissue | 66.25 (12.88) | 77.50 (18.21)
  Basal Integration: number analyzed (Participants) | 7 | 3
  Basal Integration | 82.86 (10.64) | 90.00 (16.26)
  Formation of a Tidemark: number analyzed (Participants) | 7 | 3
  Formation of a Tidemark | 65.71 (18.15) | 63.33 (27.72)
  Mid/Deep zone assessment: number analyzed (Participants) | 7 | 3
  Mid/Deep zone assessment | 50.00 (14.56) | 56.67 (22.24)
  Subcondral bone abnormalities/marrow fibrosis | 73.75 (13.45) | 77.50 (19.01)
  Surface Architecture: number analyzed (Participants) | 7 | 3
  Surface Architecture | 57.86 (11.33) | 80.00 (17.31)
  Surface/Superficial assessment: number analyzed (Participants) | 7 | 3
  Surface/Superficial assessment | 56.43 (11.42) | 83.33 (17.44)

4. Secondary Outcome: Percentage of Donor Site Refilling Based on MRI Measurements.
Description: Extent of filling of the donor site over a longer term. Percentage change from baseline in refilling of cartilage defect based on 7T MRI for donor Region.
Time Frame: Baseline, Week 4, Week 12 and Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 8 | 4
Percent
  Week 4 | 64.38 (7.80) | 38.15 (11.03)
  Week 12: number analyzed (Participants) | 7 | 4
  Week 12 | 60.25 (14.55) | 32.44 (19.09)
  Week 28 (EOS): number analyzed (Participants) | 5 | 4
  Week 28 (EOS) | 86.53 (11.09) | 62.73 (14.52)
Statistical Analysis 1: Comparison: LNA043 20mg vs Matching Placebo to 20mg; Week 4; Test type: Superiority; p = 0.0404, Mixed Effect Model Repeat Measurement; Mean Difference (Net) = 26.23, 95% CI 2-sided [-3.86 to 56.32]
Statistical Analysis 2: Comparison: LNA043 20mg vs Matching Placebo to 20mg; Week 12; Test type: Superiority; p = 0.1381, Mixed Effect Model Repeat Measurement; Mean Difference (Net) = 27.82, 95% CI 2-sided [-26.5 to 82.10]
Statistical Analysis 3: Comparison: LNA043 20mg vs Matching Placebo to 20mg; Week 28 (EOS); Test type: Superiority; p = 0.1168, Mixed Models Analysis; Mean Difference (Net) = 23.80, 96% CI 2-sided [-19.3 to 66.89]

5. Secondary Outcome: Change From Baseline in GAG Content
Description: Sodium MRI-based measurements of change from baseline in glycosaminoglycan (GAG) content was assessed from both defective sites and a nearby healthy cartilage region (as a reference tissue). Specifically, the ratio of normalized sodium signal in the surgically created defect (SCD or donor site) to healthy non-weight bearing region (HNWB), i.e. SCD/HNWB was of major interest
Time Frame: Baseline, Week 12 and Week 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 7 | 4
Ratio
  SCD/HNWB - Week 12 | 0.14 (0.07) | 0.15 (0.09)
  SCD/HNWB - Week 28: number analyzed (Participants) | 6 | 3
  SCD/HNWB - Week 28 | 0.33 (0.10) | 0.14 (0.14)
Statistical Analysis 1: Comparison: LNA043 20mg vs Matching Placebo to 20mg; SCD/HNWB - Week 12; Test type: Superiority; p = 0.5175, Mixed Effect Model Repeat Measurement; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.26 to 0.25]
Statistical Analysis 2: Comparison: LNA043 20mg vs Matching Placebo to 20mg; SCD/HNWB - Week 28; Test type: Superiority; p = 0.1476, Mixed Effect Model Repeat Measurement; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.22 to 0.60]

6. Secondary Outcome: Bi-layer Collagen Organization Based on MRI Measurements
Description: MRI T2 maps were generated and zonal T2 ratios (superficial layer T2 / deep layer T2) were calculated to assess the collagen fiber organization in the SCD cartilage region.
Time Frame: Week 12 and Week 28
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 6 | 4
Ratio
  Week 12: number analyzed (Participants) | 5 | 4
  Week 12 | 1.44 (0.15) | 1.57 (0.18)
  Week 28 | 1.33 (0.11) | 1.45 (0.14)

7. Secondary Outcome: PK Profile of LNA043 and of AngPTL3 in Serum Cmax
Description: Local and systemic pharmacokinetics (PK) of LNA043 following a single i.a. administration
Time Frame: 4 weeks
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 8 | 5
ng/mL
  LNA043: number analyzed (Participants) | 8 | 0
  LNA043 | 57.4 (22.1) |
  AngPTL3 | 22.9 (9.03) | 26.6 (7.62)

8. Secondary Outcome: PK Profile of LNA043 and of AngPTL3 in Serum AUC
Description: Local and systemic pharmacokinetics (PK) of LNA043 following a single i.a. administration
Time Frame: 4 weeks
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 8 | 5
hr*ng/mL
  LNA043: number analyzed (Participants) | 8 | 0
  LNA043 | 821 (349) |
  AngPTL3 | 3130 (1440) | 3030 (1060)

9. Secondary Outcome: Number of Participants With Anti-LNA043 Antibodies in Serum
Description: Potential immunogenicity of LNA043
Time Frame: Baseline, Week 1, Week 4, Week 12 and Week 28
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LNA043 20mg | Matching Placebo to 20mg
Number analyzed (Participants) | 9 | 5
Participants
  Day 1: anti-LNA043 antibodies present: YES | 0 | 0
  Day 1: anti-LNA043 antibodies present: NO | 9 | 5
  Day 8: anti-LNA043 antibodies present: YES | 0 | 0
  Day 8: anti-LNA043 antibodies present: NO | 9 | 5
  Day 29: anti-LNA043 antibodies present: YES | 0 | 0
  Day 29: anti-LNA043 antibodies present: NO | 9 | 5
  Day 85: anti-LNA043 antibodies present: YES | 0 | 0
  Day 85: anti-LNA043 antibodies present: NO | 9 | 5
  Day 197: anti-LNA043 antibodies present: YES | 0 | 0
  Day 197: anti-LNA043 antibodies present: NO | 9 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the dose of study treatment until up to 28 weeks post treatment
Groups:
- LNA043 20mg: LNA043 20mg
- Placebo: Placebo
Arm/Group | LNA043 20mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 4/9 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNA043 20mg (N=9) | Placebo (N=5)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Influenza like illness (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT03334812/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03334812/SAP_000.pdf